CLINICAL TRIAL: NCT07184463
Title: Chronic Pain After Thoracic Surgery: Towards a New Standard? A Comparative Prospective Study of Pain Reduction After Pulmonary Resection by VATS, RATS-OTC, and Hybrid RATS.
Brief Title: A Study of Pain Reduction After Pulmonary Resection by VATS, RATS-OTC, and Hybrid RATS.
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2026-13077
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Thoracic Surgery; Video-assisted Thoracic Surgery; Robotic-assisted Thoracic Surgery
Keywords: chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary resections surgery with three surgical approaches:: RATS-OTC (no intercostal access)
  VATS (intercostal instruments and specimen)
  RATS-TTH (intercostal instruments, out-of-cage specimen)
  Interventions: Other: Evaluation of chronic pain at 3 and 6 months after thoracic surgery

INTERVENTIONS:
Other: Evaluation of chronic pain at 3 and 6 months after thoracic surgery — The presence of persistent postoperative pain, defined as ipsilateral chest pain (on the same side as the surgery) occurring at rest and/or with coughing on a daily basis. Assessed by a 'yes' or 'no' response when asked at 3 and 6 months postoperatively.

SUMMARY:
Pulmonary resections are key in treating lung neoplasms, with techniques adapted to tumor size and location. Minimally invasive approaches like VATS have replaced open thoracotomy, but intercostal trocar placement can lead to nerve injury and chronic pain.

Robotic-assisted thoracic surgery (RATS) is usually done via a transthoracic (RATS-TT) approach using intercostal trocars. A newer "out of cage" method (RATS-OTC), using subcostal or subxiphoid ports, avoids intercostal access, potentially reducing nerve damage. A French study showed less opioid use and acute pain with RATS-OTC, but chronic pain outcomes are still unknown.

At CHUM, a hybrid RATS technique (RATS-TTH) is also used-intercostal for instruments, but with out-of-cage specimen extraction-to limit intercostal trauma.

DETAILED DESCRIPTION:
Pulmonary resections play a crucial role in the treatment of lung neoplasms, with procedures tailored to the size and location of the tumors. The minimally invasive approach, particularly via video-assisted thoracoscopic surgery (VATS), has replaced traditional thoracotomy by allowing access to the thoracic cavity through surgical trocars inserted between the ribs. However, these trocars, placed near the intercostal nerves, can cause nerve injury and chronic pain.

Robotic-assisted thoracic surgery (RATS) is typically performed via a transthoracic approach (RATS-TT), using intercostal trocars similar to those in VATS. Recently, a robotic approach known as "out of cage" (RATS-OTC) has been described, which involves the use of subcostal or subxiphoid trocar insertion. This method avoids the passage of instruments through the intercostal space, thus theoretically eliminating the risk of intercostal nerve injury. Compared to the transthoracic approach, a French team reported a reduction in opioid use and decreased intensity of acute postoperative pain with the RATS-OTC approach. However, due to the novelty of this technique, chronic pain outcomes have yet to be compared with those observed in RATS-TT or VATS.

At the CHUM, a modified transthoracic RATS technique-called the hybrid approach (RATS-TTH)-is also used. In this method, trocars are placed intercostally, but the extraction of large pulmonary specimens is performed through an out-of-cage route to minimize potential intercostal trauma related to specimen removal. Pain associated with this approach has also not been described in the literature.

Postoperative pain significantly affects recovery and long-term quality of life. Although the VATS approach reduces the severity of acute pain, chronic pain remains common and impactful. In fact, in the CRYO-VATS study conducted at CHUM between 2023 and 2025, the incidence of chronic pain following pulmonary resection via VATS (without cryoanalgesia) was 30% at 3 months and 17.5% at 6 months.

The aim of this study is to describe the incidence of chronic pain at 3 and 6 months for the three surgical approaches used at CHUM:

RATS-OTC (robotic, completely spares the intercostal space),

VATS (video-assisted thoracoscopy, with intercostal passage of instruments and pulmonary specimen),

RATS-TTH (robotic, hybrid technique with intercostal instrument passage but out-of-cage extraction of the pulmonary specimen).

The investigators hypothesize that the RATS-OTC approach will reduce the incidence of chronic pain by completely eliminating intercostal trauma. Currently, no study has reported on chronic pain outcomes comparing the RATS-TTH and RATS-OTC approaches. Simultaneous data collection from patients undergoing VATS will serve as a comparison baseline. These preliminary data will provide the foundation for a randomized controlled trial to validate the potential chronic pain benefits of these innovative surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* American Society of Anesthesiologists (ASA) score 1-3

Exclusion Criteria:

* Language barrier, psychiatric, physical or mental condition making pain assessment impossible despite prior education
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective anatomical pulmonary resection (anatomical segmentectomy, lobectomy or bilobectomy) via minimally invasive approach.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Presence of persistent postoperative pain | 3 and 6 months after surgery
  The presence of persistent postoperative pain, defined as ipsilateral chest pain (on the same side as the surgery) occurring at rest and/or with coughing on a daily basis. Assessed by a 'yes' or 'no' response when asked at 3 and 6 months postoperatively.

SECONDARY OUTCOMES:
Occurrence of a neuropathic pain component | 3 and 6 months after surgery
  The occurrence of a neuropathic pain component, assessed using the DN4-interview questionnaire, administered via telephone at 3 and 6 months to identify a neuropathic component. A score of 3 or higher is considered a positive result.
Impact of chronic pain on overall recovery | 3 and 6 months after surgery
  The impact of chronic pain on overall recovery, assessed using the Brief Pain Inventory (BPI) via telephone at 3 and 6 months. A change of 2 points or more on the 10-point pain intensity scale is considered clinically significant.
  Similarly, a change of at least 1 point on the pain interference score with quality of life is considered clinically significant.
Preoperative analgesic use | On the day of the surgery
  Preoperative analgesic use, determined by documenting the type of medication (opioids, anti-inflammatories, neuropathic pain treatments, etc.) and the dosage taken at home prior to surgery.
Overall recovery | 3 and 6 months after surgery
  Overall recovery, assessed by opioid consumption at 3 and 6 months, new prescriptions for neuropathic pain medications in the postoperative period, and whether the patient is still taking them at 3 and 6 months.
Residual pain intensity | 3 and 6 months after surgery
  Residual pain intensity, assessed using the Verbal Numerical Rating Scale (VNRS) at 3 and 6 months, on a scale from 0 to 10, where 0 represents no pain and 10 represents the worst pain imaginable.
Total length of hospital stay | On the day patient is discharged from hospital, up to two weeks
  Total length of hospital stay, measured from the end of surgery until discharge is signed.
Total opioid consumption during hospitalization | On the day patient is discharged from hospital, for an average of 1-2 days
  The total opioid consumption during hospitalization is calculated in morphine equivalents. Opioid doses will first be converted to morphine equivalents and then expressed as oral morphine equivalents (OME).
Type of chronic analgesia | 3 and 6 months after surgery
  Type of chronic analgesia used at the 3- and 6-month telephone follow-up (e.g., type and dosage of medication, transcutaneous electrical nerve stimulation (TENS), relaxation, distraction, acupuncture, and physiotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: Alex Moore, MD, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montreal, Montreal, Quebec, Canada